CLINICAL TRIAL: NCT03313349
Title: A School-Based Intervention to Improve Social Functioning in Children and Adolescents With ADHD: A Pragmatic Randomized Controlled Trial Comparing Standard and Enriched Provision.
Brief Title: A School-Based Intervention to Improve Social Functioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Behandlingsskolerne (Other)
Responsible Party: Principal Investigator, Bo Hedegaard Jacobsen, Chief Psychologist, Behandlingsskolerne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Borojonoad
Record Dates: First submitted 2017-09-11; First posted 2017-10-18 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: ADHD - Combined Type
Keywords: ADHD, Behavioral Problems, Children and Adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Problem Behavior

STUDY DESIGN:
Intervention Model Description: Design: A pragmatic RCT designed according to CONSORT guidance (CONSORT, 2010) to compare UP and ENB.
  Students, attending the schools, were randomly allocated to either UP or ENP according to a one-to-one ratio. Outcome measures (see below) were collected at pre-intervention (T1), post-intervention (T2 - 3 months post randomization) and follow up (T3 - 6 months post randomization). If possible, the a last follow up (T4 - 12 months post randomization).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants in the study are allocated to each arm by using randomization system. After determining which of the three school Units the student will attend, the participants are distributed in to one of the two arms at each school (UP & ENP).
  It is not possible to fully blind parents and students as they have to give informed consent. Teachers and social workers will be kept blind to allocation as far as possible . They are not directly involved in the treatment measured in this study, even though they play a great part in it. The blindness of the teachers and social workers is important as they will be providing the ratings used in the analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Provision (UP) (Other): Usual Provision
  Psychotherapy: 1. cognitive therapy 2.family intervention
  Interventions: Behavioral: Psychotherapy: 1. cognitive therapy 2.family intervention
- Enhanced/Need-Based Provision (ENP) (Other): Enhanced/need-based Provision
  Psychotherapy: 1.cognitive therapy 2.family intervention
  Interventions: Behavioral: Psychotherapy: 1. cognitive therapy 2.family intervention

INTERVENTIONS:
Behavioral: Psychotherapy: 1. cognitive therapy 2.family intervention — Psychotherapy delivered by trained psychologist for the student and the student´s parents

SUMMARY:
Evaluating interventions for children/adolescents with Attention Deficit Hyperactivity Disorder (ADHD) is a field that offers many challenges. Even though psychotherapeutic treatment for ADHD is recommended as the first choice in many countries(1), the evidence base for this is inconsistent and outcome specific (2). For instance, parent training may not have significant effects on the core Symptoms of ADHD (3). However, trials suggest that it facilitates skills in other areas. One area where it is of potential value is social functioning (4). The randomized controlled trial (RCT)described here will test the therapeutic value of a package of psychological interventions designed to target social functioning for children and adolescents with ADHD. It will be conducted in a special school environment designed specifically for children with severe behavioral problems. Therefore, routine provision is already substantial. As a result, it was not possible to include a "no intervention group" (control group) for ethical reasons. Therefore, the value of social skills intervention was examined by comparing different "doses" of the routine intervention by testing a usual provision (UP) group against an enriched/need-based (ENP) form of provision.

DETAILED DESCRIPTION:
Background:

In 2013, the former Danish minister of Social Affairs presented a national plan for the help and treatment of people with ADHD. Acknowledging the rise in the number of citizens in Denmark with an ADHD diagnosis, the Danish government supported an enhanced effort to offer this group adequate treatment. The government's aim was to secure an increased quality of life for individuals with ADHD.

The Ministry of Social Affairs sees ADHD as a cluster of co-occurring difficulties that creates various problems in life for affected individuals. The main goal with the national plan, was (i) to provide early years help for children, (ii) to prevent the development of ADHD type of problems, and (iii) to provide the proper treatment for people, who already have ADHD.

The plan did not consider the biological perspectives, and medicinal treatment is not mentioned as a part of the plan - while non-pharmacological interventions, such as parent training, were considered the first priority (5). This priority for non-pharmacological interventions rested partly on ethical considerations, although the report suggests that a number of training programs are evidence-based. The evidence-base for non-pharmacological interventions remains complex. For instance, the benefits of parent training and child-focused treatments for core ADHD symptom control is limited - especially when blinded outcomes are considered (6). In contrast, parent training seems to improve parenting and reduce conduct disorder (7). Social skills training may also have value (8). This is important as, although behavioral problems are not considered a core symptom in ADHD, social functioning deficits are recognized in many children with ADHD (9) and conduct disorder is a relatively common comorbidity (10).

In a society like Denmark, where people with ADHD receive psychosocial treatment and support from the Social Services before they are considered for medical treatment, it is vital that studies of nonpharmacological interventions are conducted. The investigators have to analyze to what extend the interventions can have an effect and on which areas of functioning we can expect improvement. In Denmark, children with most severe behavior problems are treated in special educational settings. In these settings, nonpharmacological treatment is the norm. Considering this, more studies should be conducted in such settings to see if the approaches used are of value.

The proposed RCT will contribute to the knowledge about the value of nonpharmacological interventions, especially with regard to social functioning and skills for ADHD, by investigating treatment in a special school setting providing care for children/adolescents with severe ADHD symptoms and behavior problems.

Aims and objectives:

The overall aim of this study is to evaluate the benefits of enriching and extending an existing non-pharmacological intervention for social skills deficits in ADHD currently delivered in a special school environment. To do this, we will compare usual provision (UP) with an enhanced and need based provision (ENP).

The main research questions are:

* Does enriching and extending an existing nonpharmacological intervention for social skills increase its effectiveness in terms of social skill improvements?
* Do these effects persist to 3, 6, and 12 months post-randomization?
* Does the enriched intervention reduce core symptoms of conduct disorder and ADHD compared to the routine one?
* Does medication taken during the study moderate the outcome?

Method:

For ethical reasons, it is not possible in this study to have a control group that does not receive treatment. The Ministry of Social Affairs legislation does not allow students to be in a control group with no treatment in a special school setting. Due to these circumstances, the study will be a pragmatic RCT study. Therefore, a two-arm RCT will be carried out to evaluate whether the effectiveness of the intervention is greater when delivered in an "enriched/need Based provision" (ENP) format compared to a "usual provision" (UP).

Study setting:

Participants will be enlisted at the three schools in Denmark; Pilelygaard, Pilen and Kompasset - each part of an organization called Behandlingsskolerne which has approximately 100 students enrolled at any time. Daily treatment is primarily offered in a school setting, but can take place elsewhere (visiting a café, walk in the park etc.). Family work will be carried out in the student´s home or at school meetings. Students in these schools do not have ASD as a primary diagnosis or a very low IQ. However, the level of comorbidity is high. More than half of the students have more than one diagnosis.

The level of staffing is high with 1:2 staff to student ratio. Many of the staff are trained to deliver psychological treatment. Both teachers and social workers are all trained in a cognitive approach and follow the guidelines of specialized psychologists in the treatment. The staff are supervised on a regular basis and participate in meetings with the school unit, class team, and the psychologists to secure every student´s progress.

Participants:

Participants in the study are all students enlisted at Behandlingsskolerne. An Organization that houses several special schools.

Inclusion criteria:

* Children from 6 to 18 years old.
* ADHD diagnosis from a psychiatric institution.
* Diagnosis F.90.1 - Hyperkinetic behavioral disorder (ICD10), or history of behavioral problems in multiple settings (School, Home, leisure time).
* Parents/caregivers with no reported mental illness or severe addictions.

Exclusion criteria:

* Pre-existing diagnosis of ASD.
* Intellectual disability with an IQ < 70 WISC.
* Pre-existing diagnosis of anxiety and/or depression.

Recruitment:

Following the Ministry of Social Affairs legislation, students with ADHD are offered private treatment in special schools when education and treatment is not possible in public schools. Each student is individually evaluated by Social Service officials before being offered private treatment. When the student´s parents and the Social Service Department first consider Behandlingsskolerne as an option, the student´s files are send to the school and a meeting is held between the parents, officials and the school. Taking into consideration the diagnosis, the school history and recommendations from the family, the student is placed in a school unit within the organization - one that is judged able to meet the student´s unique needs. The study will consider each student enlisted in these three school units between the dates 01.03.17 and 01.09.18. Students meeting the inclusion and exclusion criteria will be take part in the study.

Intervention:

The intervention in this RCT consist of two versions of a package of psychotherapeutic sessions given to the students and students' parents. Trained psychologists offer a number of sessions in which problems regarding ADHD and/or behavioral problems are addressed. The following describes the standard interventions offered at Behandlingsskolerne for children with ADHD and severe behavioral problems (The content of the therapeutic approach is available from the author):

Intervention with students:

* Therapy sessions
* Establishing relationship with student
* Psychoeducation:
* Observations
* Other

Interventions with parents:

* Therapy sessions
* Establishing relation with parents and within the family
* Psychoeducation
* Observation
* Other

The difference between the UP and ENP groups: The UP-group receives a fixed amount of intervention = five sessions (three for the student and two for the parents) each month in which relevant treatment is picked from the intervention approaches mentioned above. The ENP-group receives the same treatment options from the intervention list but in an enhanced form. This group receives not less than seven sessions (four for the student and three for the parents). Furthermore, in the ENP-Group, there is no limit regarding the number of interventions. The psychologist will evaluate how many sessions he considers are needed to progress in each case.

The psychologists will report the progress in treatment for the students in the study at monthly meetings. They track the therapy sessions offered for each student in a registration sheet. At these meetings, the ethical perspectives are discussed and the extent of the treatment is considered. If a student is not making progress, or even getting worse, a shift from the UP group to the ENP-Group is possible.

Study measures:

Diagnostic assessment:

A psychiatric assessment has been performed on every student in the study in a hospital in Denmark. These took into account the typical range of information required from an assessment from multiple sources and across multiple settings. Considering the medical history, diagnostic interviews, and test results, all students participating are diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) and not ASD or with an IQ of less than 70. Behavioral problems are diagnosed in the hospital or described in the school records.

Outcomes T1 to T4 outcomes were measured using the following scales.

Social skills (primary outcome)

* SRS - Social Responsiveness Scale - (teachers/social workers). The SRS test assess the functioning in general on five subscales: Social Cognition, Social Communication, Social Consciousness, Social Motivation, and Stereotypic behavior. The SRS is specially design to identify different types of abnormalities in social functioning and describe social problems (Wigham et al, 2012). The SRS is completed by a teacher or social worker.
* ABBAS II - Adaptive Behavior Assessment System - (for both teacher/social workers and parents). The ABAS II test assesses adaptive behavior in three domains: conceptual, social, and practical functioning. Beside the domain targeting the social skills in the test, many of the subscales can be linked to social functioning in general and the test is sensitive to progression/maturation (Harrison et al, 2003). The ABAS II is completed by both parents and teacher/social worker.

ADHD symptoms and conduct problems (secondary outcomes)

* SDQ - Strength and Difficulty Questionnaire - (teachers/social workers). The SDQ is the most used test in Denmark for screening psychopathologies. The test covers four problem areas: Hyperactivity/Attention, Behavioral Problems, Emotional Problems, and Peer Problems (Niclasen et al, 2012). The SDQ is completed by a teacher or social worker.
* ADHD-RS - Attention deficit Hyperactivity Disorder Rating Scale - (teachers/social workers). The ADHD-RS test is used to identify traits in ADHD on two subscales: Attention and Impulsivity/Hyperactivity (DuPaul et al. 1998). The ADHD-RS is completed by teacher or social worker.

Statistical analysis and sample size:

The primary analysis will employ an ITT analysis, with multiple imputation of missing data, using linear mixed models to compare the two trial arms on an aggregate score on the two social skills scales at T2. T1 scores will be included in the model as a covariate. Secondary analysis will use similar models for other outcomes at other time-points. To obtain adequate statistical power, the two treatment arms will be split equally using a 1-to-1 ratio. Clinically valuable change (MIREDIF) on the primary outcome requires a minimum 15 scale point improvement which is equivalent to a .6 standard deviation change. This require 32 Students (16 in the Study Group and 16 in the Control Group) to obtain a power of 80% (100% - errors of type II) using a conventional statistical level of significance of 5%. The group will be stratified for sex of participant and by which unit they are attending.

Moderator Analysis: We will record the nature of all treatment (including medication) received, and this will be summarized and quantified and used as a moderator in the analysis.

Ethical approval and Informed consent:

Standard ethical procedures will apply. Students and participants will give written informed consent. We are obliged to protect all data collected and the data can only be used in an anonymous form. Associate Professor Henrik Skovlund from University of Århus is responsible for monitoring and securing all the ethical aspects of the study.

Allocation and blinding:

Participants in the study are allocated to each arm by using randomization system. After determining which of the three school Units the student will attend, the participants are distributed in to one of the two arms at each school (UP & ENP).

It is not possible to fully blind parents and students as they have to give informed consent. Teachers and social workers will be kept blind to allocation as far as possible . They are not directly involved in the treatment measured in this study, even though they play a great part in it. The blindness of the teachers and social workers is important as they will be providing the ratings used in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 18 years old.
* ADHD diagnosis from a psychiatric institution.
* Diagnosis F.90.1 - Hyperkinetic behavioral disorder (ICD10), or history of behavioral problems in multiple settings (School, Home, leisure time).
* Parents/caregivers with no reported mental illness or severe addictions.

Exclusion Criteria:

* Pre-existing diagnosis of ASD.
* Intellectual disability with an IQ < 70 WISC.
* Pre-existing diagnosis of anxiety and/or depression.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Total score Adaptive Behavior Assesment System (ABASII) | 0-12 month
  Primary outcome will be an aggregate score on social and adaptive functioning from the assessment using ABASII (Adaptive Behavior Assessment System).
  The score is shown as "General Adaptive Composite" (GAC) on a scale from 60 to 140. The Mean area of GAC is found on the scale between a score 90 and 109. A GAC score from 100-140 is indicating a functionning level ranging from "better than mean" to "extremely high". A GAC score from 90-60 is indicating a functioning level ranging from "below mean" to " extremly low".
Total score Social Responsiveness Scale (SRS) | 0-12 month
  Primary outcome will be an aggregate score on social functioning from the assessment using SRS (Social Responsiveness Scale).
  The score is shown as "T-Score" on a scale from 30 to 90. A T-Score below 60 indicates normal functioning in social responsiveness. A T-score between 60 and 75 indicates difficulties in a mild to moderate level. A T-Score higher than 75 indicates severe difficulties.

SECONDARY OUTCOMES:
Subscale scores Strength and Difficulties Questionnaire (SDQ) on "behavioral difficulties", "getting along with other children" and "hyperactivity and concentration difficulties". | 0-12 month
  Secondary outcome will be using subscale scores of strength and difficulties using SDQ (Strength and Difficulties Qustionnaire).
  The SDQ has 25 items on an ordinal scale:
  1. Not true
  2. Partly true
  3. True
  Each Item is scored in a range from 0-10 indicating the level of difficulties.
Total score Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) | 0-12 month
  Secondary outcome will be a an aggregate score of ADHD symptoms and conduct disorder using ADHD-RS (Attention Deficit Hyperactivity Disorder Rating Scale).
  ADHD-RS has 26 items on an ordinal scale:
  1. Rarely/Never
  2. Sometimes
  3. Often
  4. Very often
  The score is ranging from 0- 78 indicating the level of difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Skovlund, Phd, Principal Investigator — University of Aarhus
Locations (1):
- Behandlingsskolerne, Vanløse, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen PS, Hinshaw SP, Kraemer HC, Lenora N, Newcorn JH, Abikoff HB, March JS, Arnold LE, Cantwell DP, Conners CK, Elliott GR, Greenhill LL, Hechtman L, Hoza B, Pelham WE, Severe JB, Swanson JM, Wells KC, Wigal T, Vitiello B. ADHD comorbidity findings from the MTA study: comparing comorbid subgroups. J Am Acad Child Adolesc Psychiatry. 2001 Feb;40(2):147-58. doi: 10.1097/00004583-200102000-00009. PMID 11211363
- [Background] van den Hoofdakker BJ, van der Veen-Mulders L, Sytema S, Emmelkamp PMG, Minderaa RB, Nauta MH. Effectiveness of behavioral parent training for children with ADHD in routine clinical practice: a randomized controlled study. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1263-1271. doi: 10.1097/chi.0b013e3181354bc2. PMID 17885567
- [Background] Barkley RA, Fischer M. The unique contribution of emotional impulsiveness to impairment in major life activities in hyperactive children as adults. J Am Acad Child Adolesc Psychiatry. 2010 May;49(5):503-13. doi: 10.1097/00004583-201005000-00011. PMID 20431470
- [Background] Daley D, van der Oord S, Ferrin M, Danckaerts M, Doepfner M, Cortese S, Sonuga-Barke EJ; European ADHD Guidelines Group. Behavioral interventions in attention-deficit/hyperactivity disorder: a meta-analysis of randomized controlled trials across multiple outcome domains. J Am Acad Child Adolesc Psychiatry. 2014 Aug;53(8):835-47, 847.e1-5. doi: 10.1016/j.jaac.2014.05.013. Epub 2014 Jun 26. PMID 25062591
- [Background] Gol D, Jarus T. Effect of a social skills training group on everyday activities of children with attention-deficit-hyperactivity disorder. Dev Med Child Neurol. 2005 Aug;47(8):539-45. doi: 10.1017/s0012162205001052. PMID 16108454
- [Background] DuPaul, G. J., Power, T. J., Anastopoulos, A. D., & Reid, R. (1998). ADHD Rating Scale-IV: Checklists, Norms, and Clinical Interpretation. New York: Guilford.
- [Background] Harrison, P.L., & Oakland, T. (2003), Adaptive Behavior Assessment System - Second Edition, San Antonio, TX: The Psychological Corporation)
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] MTA Cooporativ Group (1999) The Multimodal Treatment of Attention Deficit Hyperactivity Disorder Study, funded by National Institute of Mental Health. JAMA Psychiatry.
- [Background] Niclasen J, Teasdale TW, Andersen AM, Skovgaard AM, Elberling H, Obel C. Psychometric properties of the Danish Strength and Difficulties Questionnaire: the SDQ assessed for more than 70,000 raters in four different cohorts. PLoS One. 2012;7(2):e32025. doi: 10.1371/journal.pone.0032025. Epub 2012 Feb 27. PMID 22384129
- [Background] Sonuga-Barke EJ, Brandeis D, Cortese S, Daley D, Ferrin M, Holtmann M, Stevenson J, Danckaerts M, van der Oord S, Dopfner M, Dittmann RW, Simonoff E, Zuddas A, Banaschewski T, Buitelaar J, Coghill D, Hollis C, Konofal E, Lecendreux M, Wong IC, Sergeant J; European ADHD Guidelines Group. Nonpharmacological interventions for ADHD: systematic review and meta-analyses of randomized controlled trials of dietary and psychological treatments. Am J Psychiatry. 2013 Mar;170(3):275-89. doi: 10.1176/appi.ajp.2012.12070991. PMID 23360949
- [Background] Wigham S, McConachie H, Tandos J, Le Couteur AS; Gateshead Millennium Study core team. The reliability and validity of the Social Responsiveness Scale in a UK general child population. Res Dev Disabil. 2012 May-Jun;33(3):944-50. doi: 10.1016/j.ridd.2011.12.017. Epub 2012 Jan 25. PMID 22277583